CLINICAL TRIAL: NCT00072176
Title: A Phase II Study of CCI-779 in Patients With Metastatic and/or Locally Advanced Recurrent Endometrial Cancer
Brief Title: Temsirolimus in Treating Patients With Metastatic or Locally Advanced Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00649; NCI-2014-00649 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I160; CAN-NCIC-IND160; IND.160; CDR0000335543; NCIC-160 (Other: National Cancer Institute of Canada Clinical Trials Group); NCIC-160 (Other: CTEP)
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2014-03

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Cell Carcinoma; Endometrial Clear Cell Carcinoma; Endometrial Papillary Serous Carcinoma; Recurrent Endometrial Carcinoma; Stage IIIA Endometrial Carcinoma; Stage IIIB Endometrial Carcinoma; Stage IIIC Endometrial Carcinoma; Stage IVA Endometrial Carcinoma; Stage IVB Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well temsirolimus works in treating patients with endometrial cancer that has spread to other parts of the body or has spread from where it started to nearby tissue or lymph nodes and has come back after a period of time during which the cancer could not be detected. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the efficacy (response rate & duration of stable disease) of CCI-779 (temsirolimus) given intravenously (IV) weekly in patients with metastatic and/or locally advanced recurrent carcinoma of the endometrium.

II. To assess the adverse events, time to progression and response duration of CCI-779 given IV weekly in patients with metastatic and/or locally advanced recurrent carcinoma of the endometrium.

III. To correlate objective tumor response with phosphatase and tensin homolog gene (PTEN) expression in the tumor tissue obtained at diagnosis (primary tumor).

IV. To explore the relationship between objective tumor response with other molecular measures in diagnostic tumor tissue.

OUTLINE:

Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed metastatic and/or locally advanced recurrent adenocarcinoma (papillary serous, papillary, villoglandular, mucinous, clear cell), endometrioid or adenosquamous carcinoma of the endometrium, incurable by standard therapies
* Patients must have tumour tissue from their primary tumor available to assess molecular markers of CCI-779 activation (paraffin block or unstained slides)
* Presence of clinically and/or radiologically documented disease; at least one site of disease must be unidimensionally measurable as follows:

  * X-ray, physical exam >= 20 mm
  * Spiral computed tomography (CT) scan >= 10 mm
  * Non-spiral CT scan >= 20 mm
  * All radiology studies must be performed within 28 days prior to registration (within 35 days if negative)
* Patients must have a life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2
* Previous therapy:

  * Hormonal therapy:

    * Group A: One prior hormonal treatment (progestational or aromatase inhibitor) as either adjuvant therapy or for treatment of metastatic disease
    * Group B: No limit to number of prior hormonal treatments given (progestational or aromatase inhibitor) as either adjuvant therapy or for treatment of metastatic disease
    * Time since last hormone: >= 1 week since last dose of hormonal therapy (applies to both Groups)
  * Chemotherapy:

    * Group A: No prior chemotherapy
    * Group B: Patients must have had one prior regimen of chemotherapy for metastatic disease; patients must be 4 weeks since last dose of chemotherapy
  * Radiation: Patients may have had prior radiation therapy; a minimum of 28 days must have elapsed between the end of radiotherapy and registration onto the study; (exceptions may be made however, for low dose, palliative radiotherapy; patients must have recovered from any acute toxic effects from radiation prior to registration
  * Previous surgery: Previous major surgery is permitted provided that it has been at least 21 days prior to patient registration and that wound healing has occurred
* Granulocytes (absolute granulocyte count [AGC]) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Bilirubin =< upper normal limit (UNL)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x UNL
* Serum creatinine =< 1.5 x UNL or creatinine clearance >= 50 ml/min; creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft Formula
* Fasting serum cholesterol =< 9.0 mmol/L
* Fasting triglycerides =< 4.56 mmol/L
* Patient consent must be obtained according to local Institutional and/or University Human Experimentation Committee requirements; it will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) Study Coordinator that such clearance has been obtained, before the trial can commence in that centre; because of differing requirements, a standard consent form for the trial will not be provided but a sample form is given; a copy of the initial full board Research Ethics Board (REB) approval and approved consent form must be sent to the central office; the patient must sign the consent form prior to randomization or registration; please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records
* Patients must be accessible for treatment and follow-up; patients registered on this trial must be treated and followed at the participating center; this implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial; investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient registration

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for >= 5 years
* Patients must not have had prior treatment with an mammalian target of rapamycin (mTOR) inhibitor
* Uterine sarcomas (leiomyosarcoma), mixed mullerian tumours (MMT) and/or adenosarcomas
* Patients with non-measurable disease only; (please note that bone metastases are considered non-measurable)
* Pregnant or lactating women; pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with CCI-779; most patients enrolled on this trial will have had a prior hysterectomy or pelvic irradiation; however, if the patient is of childbearing potential, a urine beta-human chorionic gonadotropin (HCG) must be proved negative within 7 days prior to registration; women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with known brain metastases; (a head CT is not necessary to rule out brain metastases, unless there is clinical suspicion of central nervous system [CNS] involvement)
* Patients with serious cardiovascular illness such as myocardial infarction within 6 months prior to entry, congestive heart failure (even if medically controlled), unstable angina, active cardiomyopathy, unstable ventricular arrhythmia or uncontrolled hypertension
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CCI-779
* Patients receiving concurrent treatment with other anti-cancer therapy or other investigational agents
* Serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:

  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements
  * Active uncontrolled infection
  * Active peptic ulcer disease
  * Any other medical conditions that might be aggravated by treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-05; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — Canadian Cancer Trials Group
Locations (1):
- National Cancer Institute of Canada Clinical Trials Group, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 10 participating centers across Canada between May 2004 and June 2007.
Groups:
- Group A: Chemotherapy naive patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  temsirolimus: Given IV
  laboratory biomarker analysis: Correlative studies
- Group B: Chemotherapy treated patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  temsirolimus: Given IV
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Group A | Group B
Started | 34 | 28
Completed | 33 | 27
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 33 | 27 | 60
Age, Continuous [Median (Full Range); unit: years] | 66 [52 to 80] | 60 [41 to 81] | 63 [41 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 27 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 33 | 27 | 60

OUTCOME MEASURES:

1. Primary Outcome: Objective Clinical Response Rate
Description: Defined as proportion of patients with 30% decrease in the sum of the longest diameters of the target lesions (partial response) maintained for at least 4 weeks, or complete disappearance of disease and cancer related symptoms (complete response) and confirmed on independent radiology review.
Time Frame: Up to 5 years
Population: Patients who were evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of patients with response
Arm/Group | Group A | Group B
Number analyzed (Participants) | 29 | 25
percentage of patients with response | 13.8 [3.9 to 31.7] | 4.0 [0.1 to 10.4]

2. Primary Outcome: Progression-free Survival (Tumor Progression)
Description: Time to tumor progression or death
Time Frame: 5 years
Population: All patients who were evaluable for response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 29 | 25
months | 7.33 [3.61 to 9.86] | 3.25 [1.97 to 3.84]

ADVERSE EVENTS:
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 11/33 | 9/27
Other Adverse Events (participants affected / at risk) | 33/33 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=33) | Group B (N=27)
Limb Edema (Blood and lymphatic system disorders) | 1 | 0
Hospitalization for dehydration (Gastrointestinal disorders) | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 0
Hospitalization for spinal cord compression (Nervous system disorders) | 1 | 1
Hospitalization for hyperglycemia (Investigations) | 1 | 0
Hospitalization for bowel obstruction and enteritis (Gastrointestinal disorders) | 1 | 0
Hospitalization for chest pain (General disorders) | 1 | 0
Hospitalization for pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hospitalization for abdominal pain (General disorders) | 1 | 0
Hospitalization for hypokalemia (Investigations) | 1 | 2
Hospitalization for anorexia (Gastrointestinal disorders) | 1 | 0
Hospitalization for gastrointestinal pain (General disorders) | 1 | 0
Hospitalization for renal obstruction (Renal and urinary disorders) | 1 | 0
Hospitalization for pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hospitalization for leg pain (General disorders) | 1 | 0
Hospitalization for bowel obstruction (Gastrointestinal disorders) | 1 | 0
Hospitalization for Hyponatremia (Investigations) | 0 | 1
Hospitalization for Nausea (Gastrointestinal disorders) | 0 | 1
Hospitalization for Fatigue (General disorders) | 0 | 1
Hospitalization for Vomiting (Gastrointestinal disorders) | 0 | 2
Hospitalization for diarrhea (Gastrointestinal disorders) | 0 | 2
Hospitalization for Urosepsis (Infections and infestations) | 0 | 1
Hospitalization for Anemia (Blood and lymphatic system disorders) | 0 | 1
Hospitalization for Fistula (Gastrointestinal disorders) | 0 | 1
Thrombosis (Blood and lymphatic system disorders) | 0 | 1
Hospitalization for Impending Fracture of Lytic Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hospitalization for Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hospitalization for Ear Pain (Ear and labyrinth disorders) | 0 | 1
Hospitalization for Facial Nerve & Vocal Cord Paralysis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=33) | Group B (N=27)
Allergic reaction (Immune system disorders) | 2 | 1
Rhinitis (Immune system disorders) | 7 | 2
Supraventricular arrhythmia Atrial tachycardia (Cardiac disorders) | 2 | 0
Supraventricular arrhythmia Sinus tachycardia (Cardiac disorders) | 1 | 3
Supraventricular arrhythmia Tachycardia (Cardiac disorders) | 1 | 3
Hypertension (Cardiac disorders) | 4 | 1
Hypotension (Cardiac disorders) | 2 | 0
Cardiac General - Other (Cardiac disorders) | 2 | 1
Fatigue (General disorders) | 28 | 21
Fever (General disorders) | 6 | 3
Insomnia (General disorders) | 9 | 7
Rigors/chills (General disorders) | 5 | 4
Acne (Skin and subcutaneous tissue disorders) | 5 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 4
Bruising (Skin and subcutaneous tissue disorders) | 7 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 4
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 4
Rash (Skin and subcutaneous tissue disorders) | 16 | 13
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatology - Other (Skin and subcutaneous tissue disorders) | 4 | 3
Hot flashes (Endocrine disorders) | 1 | 2
Anorexia (Gastrointestinal disorders) | 13 | 16
Constipation (Gastrointestinal disorders) | 14 | 11
Dehydration (Gastrointestinal disorders) | 4 | 2
Diarrhea (Gastrointestinal disorders) | 9 | 14
Distension (Gastrointestinal disorders) | 6 | 1
Dry mouth (Gastrointestinal disorders) | 7 | 3
Flatulence (Gastrointestinal disorders) | 4 | 1
Heartburn (Gastrointestinal disorders) | 4 | 7
Hemorrhoids (Gastrointestinal disorders) | 2 | 0
Mucositis (clinical exam) Oral cavity (Gastrointestinal disorders) | 2 | 0
Mucositis (functional/symptomatic) Oral cavity (Gastrointestinal disorders) | 21 | 18
Nausea (Gastrointestinal disorders) | 16 | 15
Taste alteration (Gastrointestinal disorders) | 14 | 8
Vomiting (Gastrointestinal disorders) | 12 | 10
GI - Other (Gastrointestinal disorders) | 3 | 2
Hemorrhage pulmonary Nose (Blood and lymphatic system disorders) | 8 | 4
Hemorrhage, GU Urinary NOS (Blood and lymphatic system disorders) | 2 | 0
Hemorrhage, GU Vagina (Blood and lymphatic system disorders) | 3 | 1
Infection with normal ANC Lip/perioral (Infections and infestations) | 4 | 1
Infection with normal ANC Lung (Infections and infestations) | 2 | 0
Infection with normal ANC Skin (Infections and infestations) | 4 | 0
Infection with normal ANC Ungual (Infections and infestations) | 3 | 0
IInfection with normal ANC Upper airway NOS (Infections and infestations) | 2 | 1
Edema: head and neck (Blood and lymphatic system disorders) | 2 | 0
Edema: limb (Blood and lymphatic system disorders) | 19 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness Extremity-lower (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 3 | 4
Mood alteration Anxiety (Nervous system disorders) | 6 | 5
Mood alteration Depression (Nervous system disorders) | 4 | 2
Neuropathy-sensory (Nervous system disorders) | 7 | 10
Somnolence (Nervous system disorders) | 2 | 1
Neurology - Other (Nervous system disorders) | 1 | 3
Dry eye (Eye disorders) | 2 | 1
Watery eye (Eye disorders) | 2 | 0
Ocular - Other (Eye disorders) | 2 | 1
Pain Abdomen NOS (General disorders) | 20 | 14
Pain Back (General disorders) | 9 | 10
Pain Bladder (General disorders) | 5 | 4
Pain Bone (General disorders) | 2 | 3
Pain Chest wall (General disorders) | 2 | 2
Pain Chest/thorax NOS (General disorders) | 3 | 1
Pain Esophagus (General disorders) | 2 | 1
Pain Extremity-limb (General disorders) | 5 | 3
Pain Head/headache (General disorders) | 10 | 5
Pain Joint (General disorders) | 6 | 4
Pain Muscle (General disorders) | 7 | 2
Pain Neuralgia/peripheral nerve (General disorders) | 2 | 0
Pain - Other (General disorders) | 3 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 | 10
Voice changes (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Incontinence, urinary (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary frequency (Renal and urinary disorders) | 6 | 1
Urinary retention (Renal and urinary disorders) | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 3 | 5
Flu-like syndrome (General disorders) | 1 | 4
Phlebitis (Vascular disorders) | 3 | 0
hrombosis/thrombus/embolism (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less